CLINICAL TRIAL: NCT04613817
Title: Prevalence and Incidence of Antibodies Against SARS-CoV-2 in Children Measured for One Year in Belgium: a Sero-epidemiological Prospective Cohort Study
Brief Title: Sero-prevalence COVID-19 Among Belgian Children
Acronym: SeCoBelChild
Status: Completed | Type: Observational
Sponsor: Sciensano (Other Government)
Collaborators: KU Leuven (Other); McGill University (Other)
Responsible Party: Sponsor
Other Study IDs: SC_044A
Record Dates: First submitted 2020-10-30; First posted 2020-11-03 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2021-10

CONDITIONS: SARS-CoV-2; SARS-CoV Infection; Covid19
Keywords: SARS-CoV-2; COVID-19; Children; Belgium; Pandemic 2020
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Based on studies in China, Iceland, the Netherlands and Italy it seems that children are less affected by SARS-CoV-2 infections and play a lesser role in the dissemination of the SARS-CoV-2 virus. It is unclear to which extend this is due to lesser exposure or an inherent decreased susceptibility to become infected. The low reported number of cases in children can be partially explained by the lower testing rates in the pediatric population.

To get insight in the transmission of SARS-CoV-2 virus in school-aged children it is necessary to compile data on infection of SARS-CoV-2 virus in the child and (pre-)adolescent population. The main objective of this study is to determine the sero-prevalence and sero-conversion of antibodies against SARS-CoV-2 in a sample of school-aged children (primary and secondary school) in Belgium at different time points. Additionally this study will gain insight in the incidence of SARS-CoV-2, the proportion of asymptomatic infections with SARS-CoV-2 and the role of COVID-19 infection in household members. It will give us the possibility to investigate potential risk factors for infection.

The study population includes primary and secondary school children from two predefined age groups (8-9 and 13-14 years old). These two groups are chosen because studies have shown more pronounced symptoms of infection and disease depending on age and because transmission dynamics also vary by age. The study population will be recruited in all Belgian schools including Brussels-Capital, Flemish and Walloon Region (including the German speaking community).

The study is a prospective cohort study. In total there will be 3 testing points with 3 months between each point. The sample size calculation indicated the inclusion of 41 randomly selected primary and 41 secondary schools and in each school 20 randomly selected pupils of the defined age groups. Parents/legal child caregiver will complete a questionnaire at each of the testing points providing basic socio-demographic characteristics (at baseline only) and risk-behavior and health characteristics including presence of symptoms during the time since the previous testing point (at each of the testing points). The questionnaire will be completed through a secured online application during the same week as the child had the saliva sample for serological testing taken.

Saliva samples will be sent to the Sciensano laboratory for serological analysis. The child's parent/legal caregiver will be informed of the serological result.

Study data will guide the Belgian policy makers in their advices to limit circulation of SARS-CoV-2 in Belgium and more specifically in their advice on measures for school-age children. This data might also be used to guide health authorities that have to decide on vaccination strategies once a vaccine is available; to decide whether children should be included for vaccination to create herd immunity or not.

ELIGIBILITY:
Inclusion Criteria:

* Primary schools: any pupil from the 3rd grade (or from the 2nd grade if not enough participants from 3rd grade are available in the selected school) who regularly attend school and is present at school at the first testing point
* Secondary schools: any pupil from 2nd grade who regularly attend school and is present at school at the first testing point
* Prior known SARS-CoV-2 infection does not exclude participation

Exclusion Criteria:

* Pupils who refuse to have the saliva sample taken
* Being a sibling of a study participant
* No informed consent form signed by parent of legal caregiver available at the recruitment

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study population includes primary and secondary school children from two predefined age groups. These two groups are chosen because studies have shown more pronounced symptoms of infection and disease depending on age and because transmission dynamics also vary by age. Adolescents of 15 year and older will not be included as their symptom patterns resembles more disease pathology of adults. Because of pragmatic and practical reasons we will include primary school children from the 3rd grade (age 8-9) and secondary schoolchildren from the 2nd grade (age 13-14).
  The study sample will be recruited in all Belgian schools including Brussels-Capital, and the Flemish and Walloon Regions (including the German speaking community). School attendance in this age group is high in Belgium, because of this, recruitment of school-age children through schools is acceptable.
Sampling Method: Probability Sample
Enrollment: 2103 (Actual)
Dates: Start 2020-12-03 (Actual); Primary Completion 2021-12-17 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change of prevalence of antibodies against SARS-CoV-2 among Belgian children aged 8-9 years | "Month 1", "Month 4", "Month 7", "Month 9" and "Month 11"
  Change in percentage of children aged 8-9 years with specific SARS-CoV-2 IgG/IgM detected in their saliva by ELISA (positive SARS-CoV-2 serological test) among all children tested
Change of prevalence of antibodies against SARS-CoV-2 among Belgian children aged 8-9 years | "Month 1", "Month 4", "Month 7", "Month 9" and "Month 11"
  Change in the absolute numbers of children aged 8-9 years with specific SARS-CoV-2 IgG/IgM detected in their saliva by ELISA (positive SARS-CoV-2 serological test) among all children tested
Change of prevalence of antibodies against SARS-CoV-2 among Belgian children aged 13-14 years | "Month 1", "Month 4" and "Month 7"
  Change in percentage of children aged 13-14 years with specific SARS-CoV-2 IgG/IgM detected in their saliva by ELISA (positive SARS-CoV-2 serological test) among all children tested
Change of prevalence of antibodies against SARS-CoV-2 among Belgian children aged 13-14 years | "Month 1", "Month 4" and "Month 7"
  Change in the absolute numbers of children aged 13-14 years with specific SARS-CoV-2 IgG/IgM detected in their saliva by ELISA (positive SARS-CoV-2 serological test) among all children tested
Change in SARS-CoV-2 seroconversion among among Belgian children aged 8-9 years | "Month 4", "Month 7", "Month 9" and "Month 11"
  Change in the percentage of children aged 8-9 years with specific SARS-CoV-2 IgG/IgM detected in their saliva by ELISA (positive SARS-CoV-2 serological test) among all children tested at each of the study follow-up testing points that did not have a positive SARS-CoV-2 serological test before.
Change in SARS-CoV-2 seroconversion among among Belgian children aged 13-14 years | "Month 4" and "Month 7"
  Change in the percentage of children aged 13-14 years with specific SARS-CoV-2 IgG/IgM detected in their saliva by ELISA (positive SARS-CoV-2 serological test) among all children tested at each of the study follow-up testing points that did not have a positive SARS-CoV-2 serological test before.
Change in SARS-CoV-2 seroconversion among among Belgian children aged 8-9 years | "Month 4", "Month 7", "Month 9" and "Month 11"
  Change in the absolute number of children aged 8-9 years with specific SARS-CoV-2 IgG/IgM detected in their saliva by ELISA (positive SARS-CoV-2 serological test) among all children tested at each of the study follow-up testing points that did not have a positive SARS-CoV-2 serological test before.
Change in SARS-CoV-2 seroconversion among among Belgian children aged 13-14 years | "Month 4" and "Month 7"
  Change in the absolute number of children aged 13-14 years with specific SARS-CoV-2 IgG/IgM detected in their saliva by ELISA (positive SARS-CoV-2 serological test) among all children tested at each of the study follow-up testing points that did not have a positive SARS-CoV-2 serological test before.

SECONDARY OUTCOMES:
Potential risk factors for the infection | "Month 1", "Month 4", "Month 7", "Month 9" and "Month 11"
  Proportion (%) infected children by probable exposure (probable or confirmed COVID-19 case in family or school), risk behavior and by health characteristics (co-morbidities, presence of symptoms, use of medications).
The proportion of asymptomatic cases among new cases that develop during a period of 7 months | "Month 1", "Month 4", "Month 7", "Month 9" and "Month 11"
  Percentage of asymptomatic cases among new cases (positive serological test) that develop during a period of 7 months
The proportion of asymptomatic cases among new cases that develop during a period of 7 months | "Month 1", "Month 4", "Month 7", "Month 9" and "Month 11"
  Absolute number of asymptomatic cases among new cases (positive serological test) that develop during a period of 7 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sciensano, Brussels, Belgium

REFERENCES:
- [Derived] Callies M, Kabouche I, Desombere I, Merckx J, Roelants M, Vermeulen M, Duysburgh E. SARS-CoV-2 infection prevention and control measures in Belgian schools between December 2020 and June 2021 and their association with seroprevalence: a cross-sectional analysis of a prospective cohort study. BMC Public Health. 2023 May 16;23(1):898. doi: 10.1186/s12889-023-15806-5. PMID 37194008